CLINICAL TRIAL: NCT05823597
Title: Effects of a Novel Intervention to Reduce Dietary Added-Sugar Consumption During the Transition to College: A Cluster Randomized Controlled Trial
Brief Title: Reducing Dietary Added-Sugar Consumption During the Transition to College
Acronym: ASUsugarLIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ASU SugarStudy LIA101
Record Dates: First submitted 2023-03-27; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Dietary Added Sugar Consumption
Keywords: added sugar; eating behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial
Who Masked: Participant
Masking Description: Participants were unaware that another condition existed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugar Intensive Treatment (Experimental): The Sugar-Intensive Intervention touched on exercise, sleep, and other aspects of healthy diet, but focused primarily on added sugar reduction. Beyond defining added sugar, the sugar-intensive intervention also included: information on how sugar is metabolized; description of health risks associated with excessive added sugar; opportunities to rehearse women's and men's recommended daily maxima; a game guessing the sugar content of various foods and beverages; information on proportion of undergraduates at their university who report being motivated to reduce their sugar intake; training in finding added-sugar information in nutritional labels; and concrete suggestions for replacing high-sugar foods and beverages with healthy options, and managing tempting situations.
  Interventions: Behavioral: Sugar Intensive Treatment
- General Health Control (Active Comparator): The General Health Intervention presentation covered Healthy People 2030 goals regarding physical activity (aerobic exercise, strength training), healthy eating (fruit, vegetable, and whole grain consumption; decreasing consumption of saturated fats and added sugar), and sleep (minimum of 7 hours per night), as well as healthy stress management/emotion regulation. The health benefits/risks associated with each goal were described, along with suggested strategies for achieving each goal. This version of the intervention also included a definition of added sugar and information about the recommended daily added-sugar maxima for women and men, but served mainly as an active control condition for testing the effects of the target intervention of interest.
  Interventions: Behavioral: General Health Control

INTERVENTIONS:
Behavioral: Sugar Intensive Treatment — see arm description
  Arms: Sugar Intensive Treatment
Behavioral: General Health Control — see arm description
  Arms: General Health Control

SUMMARY:
The goal of this cluster randomized controlled trial was to compare the effects of two single-session interventions (sugar-intensive vs. general health control) on added sugar intake, motivation to reduce sugar consumption, and factual knowledge about added sugar 6 weeks later, in a sample of first-semester undergraduates.

DETAILED DESCRIPTION:
Excessive sugar consumption is recognized as a critical public health concern. For many young adults, the transition to college presents both risk and a promising opportunity to encourage formation of healthy dietary habits. Capitalizing on this window of opportunity, we conducted a cluster-randomized controlled trial to compare the effects of two single-session interventions on added sugar intake in a sample of first-semester undergraduates. Participants received either an intervention primarily focused on reducing added sugar consumption or a general health behavior intervention with units on physical activity, sleep, and healthy diet. Participants' added sugar intake, motivation to reduce sugar consumption, and factual knowledge about added sugar intake were compared at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Students aged 18 years and older, enrolled in online sections of a required transition-to-college course at a large public university in the Southwest region of the U.S. All students in online sections of this class received the single-session intervention during their normal class period, early in the Fall 2020 semester, and were eligible to participate.

Exclusion Criteria:

* Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Added-Sugar Consumption at 6 Weeks | 6 weeks post-intervention
  Change from baseline in consumption of specific high-sugar foods and beverages each day during the week preceding assessment. Using a matrix with days as columns and food/beverage items as rows, participants reported number of servings consumed of each food per day of that week: regular soda/pop/sweet iced tea (12oz), energy drinks (1 can), fully sweetened sports drinks (12oz), sugar-syrup coffee drinks (small = 8-12 oz = 1 serving; med = 1.5 servings; large = 2 servings), mixed drinks/cocktails (1 drink), donut/sweet pastry/danish (1 whole), muffin/cake-type bread slice (1 whole), fresh flavored yogurt (½ cup), cookie/brownie (3 oz), cupcake/slice of cake (1 whole), slice of pie (1 whole), ice cream/frozen yogurt (½ cup), and candy (¼ cup). Servings were multiplied by grams added sugar/serving for each item based on the National Cancer Institute Dietary Health Questionnaire-III, and summed across items to obtain total weekly added sugar.

SECONDARY OUTCOMES:
Motivation to reduce added-sugar consumption | 6 weeks post-intervention
  "How motivated are you to reduce your added-sugar consumption?" Response options were 1 = Not at all motivated, 2 = A little motivated, 3 = Somewhat motivated, and 4 = Very motivated.
Added sugar factual knowledge | 6 weeks post-intervention
  Participants' knowledge of factual information regarding added sugar was assessed through three sets of questions. The first set of knowledge checks included eight statements about added sugar that participants marked as true or false (e.g., "Glucose is the primary fuel used by the human body"); the number of correct answers was summed. Second, participants were presented with a list of 12 ingredients (e.g., aspartame, honey, stevia) and asked to report whether each ingredient counts as added sugar; again, number of correct answers was summed. Third, participants were asked to state the maximum grams of added sugar per day recommended by the American Heart Association, separately for women and men, as presented in the intervention.
Change from Baseline Sleep at 6 Weeks | 6 weeks post-intervention
  Participants indicated the amount of sleep they got, in hours, for each of the last seven nights. Participants were presented with seven text boxes labeled "7 days ago", "6 days ago" … "Last night," and asked to fill in the number of hours slept for each. Responses were averaged to obtain a single hours/night score.
Change from Baseline Exercise at 6 Weeks | 6 weeks post-intervention
  Exercise was defined for participants as "any physical activity that gets the heart working much faster, makes you break a sweat, and/or requires a lot of muscle effort." Participants indicated the amount of exercise they got for each of the last seven days; response options for each day were: "none", "15 minutes", "30 minutes", "45 minutes", "60 minutes", and "more than 60 minutes." Responses were averaged to obtain a single minutes/day score.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data, study protocol, and analytic code will be made publicly available via OSF upon acceptance of the first manuscript for publication.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Upon acceptance of the initial manuscript reporting study results for publication; permanently